CLINICAL TRIAL: NCT01957384
Title: An Open-labelled, Randomized, Controlled, Comparative, Single Country (Denmark), Explorative, Cross-over Study Investigating the Performance and Safety of New 1-piece Open Ostomy Appliances Compared to Standard Care 1-piece Open Ostomy Appliances in 25 Subjects With Ileostomy
Brief Title: Investigation of the Performance and Safety of New 1-piece Open Ostomy Appliances Compared to Standard Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CP221
Record Dates: First submitted 2013-02-22; First posted 2013-10-08 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1; First Coloplast Test product 1 (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Coloplast Test product 1 are randomised to secondly test either:
  1. Coloplast Test product 2 and thereafter Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)
  2. Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)and thereafter Coloplast Test product 2
  Interventions: Device: Coloplast Test product 1; Device: Coloplast Test product 2; Device: Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)
- Treatment 2; First Coloplast Test product 2. (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Coloplast Test product 2 are randomised to secondly test either:
  1. Coloplast Test product 1 and thereafter Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)
  2. Standard Care Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)and thereafter Coloplast Test product 1
  Interventions: Device: Coloplast Test product 1; Device: Coloplast Test product 2; Device: Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)
- Treatment 3,First Standard care (see below) (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Standard Care Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active) are randomised to secondly test either:
  1. Coloplast Test product 1 and thereafter Coloplast Test product 2
  2. Coloplast Test product 2 and thereafter Coloplast Test product 1
  Interventions: Device: Coloplast Test product 1; Device: Coloplast Test product 2; Device: Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)

INTERVENTIONS:
Device: Coloplast Test product 1 — Coloplast Test product 1 is a new ostomy appliance developed by Coloplast.
Device: Coloplast Test product 2 — Coloplast Test product 2 is a new ostmoy appliance developed by Coloplast A/S
Device: Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active) — Standard Care was the subject usual ostomy appliance and had to be one of the following:
  * Coloplast: SenSura, 1-piece open bag without inspection window, size midi and maxi, custom-cut,
  * Dansac: Nova 1 & Nova Life, 1-piece open bag, size midi and maxi, custom-cut baseplate
  * Hollister: Moderma Flex, 1-piece open, size midi and maxi, custom-cut baseplate
  * ConvaTec: Esteem, 1-piece open bag, size midi and maxi, custom-cut baseplate
  * B. Braun: Flexima Active & Softima, 1-piece open bag, size midi and maxi, custom-cut baseplate

SUMMARY:
To assess the functionality and safety of the test products and also assess the products' ability to collect stool without interfering with the stoma. The degree of leakage using the product will also be measured

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Be at least 18 years of age and have full legal capacity
* Be able to handle the bags themselves or with help from caregiver
* Have an ileostomy with a diameter between 15 and 45 mm
* Have had their ostomy for at least three months
* Currently use a 1-piece flat standard care product with open bag
* Negative result of a pregnancy test for women of childbearing age
* Custom-cut product user
* Be suitable for participation in the investigation

Exclusion Criteria:

* Use irrigation during the study (flush the stoma with water)
* Currently receiving or have within the past 2 months received radio- and/or chemotherapy
* Currently receiving or have within the past month received local or systemic steroid treatment in the peristomal area
* Are pregnant or breastfeeding
* Participating in other interventional clinical investigations or have previously participated in this investigation
* Max three days wear time
* Suffer from peristomal skin problems that preclude participation in the investigation (assessed by the investigation nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte Petersen, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited through the Coloplast database in Denmark
Pre-assignment Details: 25 subjects signed informed consent and were randomized. 2 subjects were screening failures and did not test any products. One subject violated an inclusion criterion (convex user). The subject tested both test products and is therefore included in the safety population.
  The 3 subjects are not included in the participant flow below.
Groups:
- First Test Product 1, Then Test Product 2;Then Standard Care: The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Coloplast Test product 1 are randomised to secondly test :
  - Coloplast Test product 2
  and thereafter
  - Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)and thereafter Coloplast Test product 2
- First Test Product 1, Then Standard Care, Then Test Product 2: The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Coloplast Test product 1 are randomised to secondly test :
  1) Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)
  and thereafter
  1) Coloplast Test product 2
- First Test Product 2, Then Test Product 1, Then Standard Care: The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Coloplast Test product 2 are randomised to secondly test
  1) Coloplast Test product 1
  and thereafter
  1) Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)
- First Test Product 2; Then Standard Care, Then Test Product 1: The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Coloplast Test product 2 are randomised to secondly test :
  1) Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)
  and thereafter
  1) Coloplast Test product 1
- First Standard Care, Then Test Product 1, Then Test Product 2: The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)are randomised to secondly test
  1) Coloplast Test product 1
  and thereafter
  1) Coloplast Test product 2
- First Standard Care, Then Test Product 2, Then Test Product 1: The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects first testing Standard Care (Coloplast SenSura; Dansac Nova 1; Hollister Moderma FLex; Convatec Esteem; B.Braun Flexima Active)are randomised to secondly test
  1) Coloplast Test product 2
  and thereafter
  1) Coloplast Test product 1
Period: Test Period 1 (14 Days)
Arm/Group | First Test Product 1, Then Test Product 2;Then Standard Care | First Test Product 1, Then Standard Care, Then Test Product 2 | First Test Product 2, Then Test Product 1, Then Standard Care | First Test Product 2; Then Standard Care, Then Test Product 1 | First Standard Care, Then Test Product 1, Then Test Product 2 | First Standard Care, Then Test Product 2, Then Test Product 1
Started | 4 | 4 | 4 | 4 | 3 | 3
Completed | 4 | 4 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Period 2 (14 Days)
Arm/Group | First Test Product 1, Then Test Product 2;Then Standard Care | First Test Product 1, Then Standard Care, Then Test Product 2 | First Test Product 2, Then Test Product 1, Then Standard Care | First Test Product 2; Then Standard Care, Then Test Product 1 | First Standard Care, Then Test Product 1, Then Test Product 2 | First Standard Care, Then Test Product 2, Then Test Product 1
Started | 4 | 4 | 4 | 4 | 3 | 3
Completed | 4 | 4 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Period 3 (14 Days)
Arm/Group | First Test Product 1, Then Test Product 2;Then Standard Care | First Test Product 1, Then Standard Care, Then Test Product 2 | First Test Product 2, Then Test Product 1, Then Standard Care | First Test Product 2; Then Standard Care, Then Test Product 1 | First Standard Care, Then Test Product 1, Then Test Product 2 | First Standard Care, Then Test Product 2, Then Test Product 1
Started | 4 | 4 | 4 | 4 | 3 | 3
Completed | 4 | 4 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two subjects were screening failiures and did not test any test product, but did contribute with baseline data. These subjects are not inclæuded in the participant flow (as the did not test products) but contributed with baseline data.
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage was measured on a 24-point scale 0 (best possible outcome) to 24 (worst possible outcome) developed by Coloplast A/S
Time Frame: Up to 14 days per test product
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Coloplast Test Product 1: leakage data from all Test 1 baseplates
- Coloplast Test Product 2: Leakage data from all Test 2 baseplates
- Standard Care: leakage data from all Standard Care baseplates
Arm/Group | Coloplast Test Product 1 | Coloplast Test Product 2 | Standard Care
Number analyzed (Participants) | 22 | 22 | 22
Number analyzed (baseplates) | 148 | 152 | 66
units on a scale | 4 (5) | 4.6 (5.6) | 2.6 (3.7)

ADVERSE EVENTS:
Groups:
- Coloplast Test Product 1: data from all subjects who tested Test 1 baseplates
- Coloplast Test Product 2: data from all subjects who tested Test 2 baseplates
- Standard Care: data from all subjects who tested Standard Care baseplates
Arm/Group | Coloplast Test Product 1 | Coloplast Test Product 2 | Standard Care
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 5/22 | 6/22 | 3/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product 1 (N=22) | Coloplast Test Product 2 (N=22) | Standard Care (N=22)
Gastroenterit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to the test product
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product 1 (N=22) | Coloplast Test Product 2 (N=22) | Standard Care (N=22)
Peristomal skin problem (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) — Related to the test products
Bleeding from stoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Related to the test products
respirational tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Not related to the test products
infection of the operational wound on the back/ haemtom in operational wound (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — not related to the test products
Diarre (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) — not related to the test products
inflammation in rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — not related to the test products
Pain in collapsed forefoot (General disorders) | 0 (0) | 0 (0) | 1 (1) — Not relate to the test products
Gastroenterit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the test products
short term dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to test product
stinging skin around the stoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — not related to the test products

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes